CLINICAL TRIAL: NCT03154853
Title: Neuromuscular Assessments of Foot Intrinsic Muscles: (1) Between Individuals With and Without Functional Flatfoot and (2) Before and After a 3-week Short Foot Exercise Training in Individuals With Functional Flatfoot
Brief Title: Neuromuscular Study to Assess Foot Intrinsic Muscles
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 201607074RINB
Record Dates: First submitted 2017-05-08; First posted 2017-05-16 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Flexible Flatfoot
Keywords: Electromyography,Excessive Foot Pronation,exercise,neurology,physical therapy
MeSH Terms: conditions — Flatfoot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- normal foot (No Intervention): no intervention
- functional flatfoot (Experimental): Behavioral: short foot exercise
  Interventions: Other: Behavioral: short foot exercise

INTERVENTIONS:
Other: Behavioral: short foot exercise — Behavioral: short foot exercise 30 repetitions per section (10 seconds for each contraction, 1 minute between sections), 3 times/ week, 3 weeks
  Arms: functional flatfoot

SUMMARY:
The purposes of these studies are to investigate:

Differences in abductor hallucis muscles'EMG activities during different postural tasks between individuals with normal foot alignment and functional flat foot. Differences in abductor hallucis muscles'H-reflex amplitudes between individuals with normal foot alignment and functional flat foot. Changes in abductor hallucis muscles'EMG activities during different postural tasks after a 3-week short foot exercises training regimen in individuals with functional flat foot. Changes in abductor hallucis muscles'H-reflex amplitudes after a 3-week short foot exercises training regimen in individuals with functional flat foot. hypotheses: Peak-to-peak amplitudes and ratios of abductor hallucis muscles and tibialis anterior muscles during different postural tasks were significantly lower in individual with functional flat foot when compared to those with normal foot alignments. H-reflex amplitudes of abductor hallucis muscles were significantly lower in individual with functional flat foot when compared to those with normal foot alignments. Changes of peak-to-peak amplitudes and ratios of abductor hallucis muscles and tibialis anterior muscles during different postural tasks were significantly different in individuals with functional flat foot after a 3-week short foot exercise training regimen. Changes of H-reflex amplitudes of abductor hallucis muscles were significantly different in individuals with functional flat foot after a 3-week short foot exercise training regimen

ELIGIBILITY:
: Inclusion Criteria:

* Age between 20 and 45 years
* No ankle injury within the previous 6 months
* No diagnosed lower extremity injuries
* No ankle pain at the time of the study
* Foot posture index score: 0 to +5 for the normal foot (NF) group; +6 to +12 for the functional flat foot (FFF) group
* Navicular drop: 5-9 mm for the NF group; > 10 mm for the FFF group

Exclusion Criteria:

* Foot posture index score: <0
* Navicular drop< 5 mm
* Leg length discrepancy > 1.5 cm
* Diagnosed severe scoliosis
* Neurological injuries over lower extremities

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2016-11-04 (Actual); Primary Completion 2017-09-30 (Estimated); Study Completion 2017-12-30 (Estimated)

PRIMARY OUTCOMES:
Muscle activities: EMGs (mV) | Baseline
  EMGs (mV) in each posture
Muscle activities: H-reflexes (mV) | Baseline
  H-reflexes (mV) in each posture
Muscle activities change will being assessed: EMGs (mV) | Baseline. week 3
  EMGs (mV) in each posture
Muscle activities change will being assessed: H-reflexes (mV) | Baseline. week 3
  H-reflexes (mV) in each posture

CONTACTS AND LOCATIONS:
Overall Officials: Jen Yu Chen, Study Chair — School and Graduate Institute of Physical Therapy of National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No